CLINICAL TRIAL: NCT03468400
Title: Evaluation of the Reliability and Validity of a Diagnostic Sleep Disorders Questionnaire
Status: Completed | Type: Observational
Sponsor: Dayzz Live Well Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Dayzz
Record Dates: First submitted 2018-03-12; First posted 2018-03-16 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Sleep Apnea Syndromes; Insomnia; Insufficient Sleep Syndrome; Circadian Rhythm Disorders
Keywords: sleep disorders; assessment; diagnosis
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders; Sleep Deprivation; Chronobiology Disorders; Sleep Wake Disorders; Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to develop and test a user-friendly, accessible approach to sleep assessment which can function as an initial "triage" of targeted sleep conditions, such as insomnia, insufficient sleep syndrome, sleep apnea syndromes/snoring, and circadian sleep/wake disorders, within the clinical and community population. Specifically, this study will test the validity and reliability of a self-rated, digitized, and cost-effective diagnostic measure with sufficient sensitivity to accurately assess/diagnose common sleep conditions and/or risk for these conditions. Such an approach, would allow for faster assessment of common sleep conditions and disorders, and provide clinical knowledge to the individual, the physician, and if required insurance companies, as to those persons who need more immediate attention or treatment for their sleep condition.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 21-65 years who are referred to the sleep clinic at Carmel Medical Center and who are capable of filling out an electronic questionnaire in Hebrew.

Exclusion Criteria:

1. Patient age <21 years or >65 years.
2. Women who are pregnant or breastfeeding.
3. Nighttime shift-workers.
4. Persons who are unable to provide consent due to mental incapacity.
5. Persons referred for evaluation by Ministry of Transportation (for licensing purposes).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A general community population and clinical population physician-referred for diagnosis and assessment of sleep disorders at a sleep clinic within a large medical center.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Sleep disorders diagnosis and severity of diagosis | 30-60 minutes
  Dayzz diagnostic sleep questionnaire (dDSQ): Insomnia, insufficient sleep syndrome, circadian sleep/wake disorders, risk for sleep apnea, snoring

CONTACTS AND LOCATIONS:
Locations (2):
- John Hopkins University, Baltimore, Maryland, United States
- Carmel Hospital, Haifa, Israel